CLINICAL TRIAL: NCT03321162
Title: Accuracy of Guided Implant Placement Using Double Versus Triple Scan Protocol in Completely Edentulous Patients : Randomized Clinical Trial
Brief Title: Accuracy of Guided Implant Placement Using Double Versus Triple Scan Protocol in Completely Edentulous Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa mohamed el maghraby, principal investigator, Cairo University
Other Study IDs: Cebc.cu. cairo university
Record Dates: First submitted 2017-10-22; First posted 2017-10-25 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Dental Implantation
Keywords: surgical guide , double scan , triple scan protocol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- double scan protocol: In C1(double scan technique) , after CT scan for patient wearing scan appliance , two optical scan for the model with and without scan appliance.
- triple scan protocol: In C2 (triple scan technique) , after CT scan for patient wearing scan appliance , CT scan for scan appliance alone .
  Interventions: Diagnostic Test: scan protocol

INTERVENTIONS:
Diagnostic Test: scan protocol — Scanning strategy is based on multiple scans. Essentially one CT scan of the patient (usually with a scan appliance). Another CT scan of the model or scan appliance may be required (double scan technique). Such a second CT scan can be replaced by optical scanning of the model and scan appliance (triple scan technique).
  Groups: triple scan protocol

SUMMARY:
16 implant placement by surgical guide using double scan protocol versus triple scan protocol to Evaluate angular and linear deviation of virtual implants and actual implant position in completely edentulous patients according to scanning protocol C1(double scan technique) and C2 (triple scan technique) .

DETAILED DESCRIPTION:
In this study we discuss linear and angular deviation of actual implant position using planning protocol C1(double scan technique) or C2 (triple scan technique) in completely edentulous patient .

Both protocols C1(double scan technique) and C2 (triple scan technique) indicated in completely edentulous patient and require C.T scan for patient wearing scan appliance .

In C1(double scan technique) , after CT scan for patient wearing scan appliance , two optical scan for the model with and without scan appliance.

In C2 (triple scan technique) , after CT scan for patient wearing scan appliance , CT scan for scan appliance alone .

Teeth positions in both protocols were identified by radio-opaque scan appliance .

16 implant placement by surgical guide using double scan protocol versus triple scan protocol ( two groups - 8 implants in each group ) to Evaluate angular and linear deviation of virtual implants and actual implant position in completely edentulous patients according to scanning protocol C1(double scan technique) and C2 (triple scan technique) .

ELIGIBILITY:
Inclusion Criteria:

1. patients totally edentulous arches.
2. patients with Bucco-lingual bone thickness >6 mm allowing flapless implant placement
3. patients free from any systemic diseases that may affect bone quality e.g diabetes.

Exclusion Criteria:

1. patients with thin ridges.
2. patients with systemic disease that may affect bone quality.
3. Patients with poor oral hygiene and active periodontal diseases.
4. Anatomical situations requiring regenerative procedure.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients receiving dental implants in both arches by guided surgery using double versus triple scan protocol .
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2017-11-20 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of angular deviation between planned implants in surgical guide and actual implant position in completely edentulous patients . | immediate post operative
  Evaluation of angular deviation between planned implants in surgical guide and actual implant position in completely edentulous patients according to scanning protocol C1(double scan technique) and C2 (triple scan technique) .

SECONDARY OUTCOMES:
Evaluation of linear deviation between planned implants in surgical guide and actual implant position in completely edentulous patients | immediate post operative
  Evaluation of linear deviation between planned implants in surgical guide and actual implant position in completely edentulous patients according to scanning protocol C1(double scan technique) and C2 (triple scan technique) .